CLINICAL TRIAL: NCT03910309
Title: A Prospective Investigation Comparing Bone Graft Extenders in Transforaminal Interbody Fusions (TLIF) With an Acid Etched Titanium Implant: A Clinical Outcomes and Cost Analysis
Brief Title: Titan Spine Endoskeleton TT/TO Study
Status: Terminated | Type: Observational
Sponsor: Titan Spine (Industry)
Responsible Party: Sponsor
Other Study IDs: TLIF1-150
Record Dates: First submitted 2016-08-15; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Degenerative Disc Disease, Spondylolisthesis
Keywords: degenerative disc disease, spondylolisthesis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1 or 2 level TLIF candidates: Any subject determined to ALREADY be a candidate for 1 or 2 level transforaminal interbody fusion surgery
  Interventions: Device: TLIF with Titan TT/TO interbody cage

INTERVENTIONS:
Device: TLIF with Titan TT/TO interbody cage — fusion surgery

SUMMARY:
This is a prospective, multi-center controlled observational clinical study. All subjects will receive Titan Endoskeleton TT/TO acid etched titanium implant for the planned procedure. Each site will have a predetermined bonegraft extender to be used in all enrolled subjects at that site.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18-75 years of age, and skeletally mature
2. Have clinical and radiological evidence of degenerative disc disease at one or two levels of the lumbar spine between L2-S1. May also have spondylosis, spinal stenosis, or spondylolisthesis at these levels.
3. In the opinion of the treating surgeon, must already be a qualified candidate for lumbar fusion surgery including 6 months of conservative care prior to surgical intervention.
4. Psychosocially, mentally and physically able to comply with protocol, post-operative management and follow-up schedule.
5. Subject must understand and sign the written Informed Consent.

Exclusion Criteria:

1. Previous history of fusion surgery at the index level(s).
2. Clinical, laboratory and/or radiological evidence of back pain secondary to acute or chronic infection, malignancy, other space occupying lesions and metabolic bone demineralization diseases (e.g. osteomalacia, gout, Paget's disease etc.)
3. Osteoporosis defined as a DEXA bone density measurement T score ≤ 2.5 (Necessity for DEXA scan will be determined by investigator's standard of care)
4. Any terminal or autoimmune disease including but not limited to HIV infection, rheumatoid arthritis or lupus.
5. Any other concurrent medical disease that might impair normal healing process.
6. Morbid obesity (BMI ≥ 40 kg/m2).
7. Investigational drug or device use within 30 days.
8. Currently a prisoner.
9. Currently experiencing a major mental illness (psychosis, schizophrenia, major affective disorder) which may indicate that the symptoms are psychological rather than of physical origin.

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred and fifty (150) subjects will participate in the study at a max of 15 clinical sites. All subjects will have been diagnosed with lumbar spine disease at one or two levels of the lumbar spine that requires lumbar interbody fusion procedure as per the opinion of the treating surgeon.Subjects will be offered the opportunity to participate in the trial if he/she is determined to be a candidate for TLIF fusion surgery. The population will be drawn from an existing patient population per participating site.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-01; Primary Completion 2018-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Pain measured by VAS | 2 years
  1 to 10
Function measured by oswestry disability index | 2 years
  10 question score

SECONDARY OUTCOMES:
Success of fusion | 3 months, 6 months, 12 months, 24 months
  Fusion will be assessed by AP/Lat Flex/Ext radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Reginald Davis, MD, Principal Investigator — Laser Spine Institute
Locations (8):
- United States (8):
  - Kenai Spine, Soldotna, Alaska
  - Spine Care Institute, Daly City, California
  - Spine Clinic of Monteray bay, Soquel, California
  - Laser Spine Institute, Tampa, Florida
  - Polaris Spine, Atlanta, Georgia
  - Chatham Orthopedic Associates, Savannah, Georgia
  - Spine Institute of Idaho, Meridian, Idaho
  - Southern Oregon Orthopedics, Medford, Oregon